CLINICAL TRIAL: NCT05213026
Title: Effects of Apexification and Regenerative Endodontic Therapy on the Periapical Bone in Immature Teeth: a Retrospective Study
Brief Title: Comparison of Apexification and Regenerative Endodontic Therapy: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Istanbul Kent University (Other); Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Assoc. Prof., Istanbul University
Other Study IDs: 2019/53
Record Dates: First submitted 2022-01-18; First posted 2022-01-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Regenerative Endodontic; Apexification; Fractals
MeSH Terms: interventions — Regenerative Endodontics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Apexification: Apexification treatment was applied by a single operator (GK) in Istanbul University Faculty of Dentistry, Department of Pedodontics,
  * Having no systemic or periodontal problems,
  * Asymptomatic or diagnosed with apical periodontitis with fistula tract,
  * Not having external/internal resorption, fracture, more than one root/canal,
  * Root canal filling is sufficient for the MTA,
  * Root canal filling and coronal restorations were completed in Istanbul University Faculty of Dentistry Department of Pedodontics,
  * Cases with periapical radiographs taken before the procedure and at least one year after the procedure was included.
- Regenerative: Apexification treatment was applied by a single operator (GK) in Istanbul University Faculty of Dentistry, Department of Pedodontics,
  * Having no systemic or periodontal problems,
  * Asymptomatic or diagnosed with apical periodontitis with fistula tract,
  * Not having external/internal resorption, fracture, more than one root/canal,
  * Root canal filling and coronal restorations were completed in Istanbul University Faculty of Dentistry Department of Pedodontics,
  * Cases with periapical radiographs taken before the procedure and at least one year after the procedure was included.
  Interventions: Procedure: Regenerative endodontics

INTERVENTIONS:
Procedure: Regenerative endodontics — Regenerative endodontic procedure with 3 Mix-MP
  Groups: Regenerative

SUMMARY:
In this study, the effects of mineral trioxide aggregation (MTA) apexification and regenerative endodontic treatment (RET) methods on periapical healing was compared with fractal analysis (FD) and periapical index (PAI).

DETAILED DESCRIPTION:
The fractal dimension analysis of each radiograph was performed using the box-counting method proposed by White and Rudolph [1] (Figure 1). All periapical radiographs in high resolution Jpeg format to be included in the study was converted to tagged image file formats (TIFF). Each ROI at 18 x 19 pixels and 2 mm from the radiographic apex was selected, cropped and amplified. "Gaussian Blur" was used to eliminate the brightness changes due to soft tissues and variable bone thicknesses. The resulting image was then be subtracted from the original image. Bone marrow spaces and trabeculae were separated from each other by adding 128 gray values to each pixel location. The fractal dimension was calculated after the binary, etching, dilate, inversion and skeletonization operations were done.

This study was carried out on the radiographic records of patients who applied to Istanbul University Faculty of Dentistry, Department of Pedodontics, who had at least one immature incisor treated with MTA apexification and RET method, and who had at least one-year follow-up radiographs.

Cases in which all endodontic treatments were performed by the same pedodontist (GK) were examined.

ELIGIBILITY:
Inclusion Criteria:

* Apexification treatment was applied by a single operator (GK) in Istanbul University Faculty of Dentistry, Department of Pedodontics,

  * Having no systemic or periodontal problems,
  * Asymptomatic or diagnosed with apical periodontitis with fistula tract,
  * Not having external/internal resorption, fracture, more than one root/canal,
  * Root canal filling is sufficient for the MTA group,
  * Root canal filling and coronal restorations were completed in Istanbul University Faculty of Dentistry Department of Pedodontics,
  * Cases with periapical radiographs taken before the procedure and at least one year after the procedure was included.

Exclusion Criteria:

* Cases treated by different pediatric dentists,

  * Cases in which apexification is performed by different operators,
  * Cases with systemic or periodontal disease,
  * Cases with external/internal resorption, fracture, more than one root/canal,
  * Cases where root canal filling is not sufficient
  * Cases in which root canal filling and conoral restorations were completed over 2 years,
  * Cases without radiographs taken before or at least one year after the procedure,
  * Cases with artifacts in the periapical region on their radiographs

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The database of patients who underwent apexification treatment by a single operator (GK) at Istanbul University Faculty of Dentistry, Department of Pedodontics was examined.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Healing | 1 year
  PAI score ≤ 3

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No